CLINICAL TRIAL: NCT03378089
Title: The Effects of Pre-Transplant Music Therapy for Patients Undergoing Hematopoietic Stem Cell Transplant
Brief Title: Music Therapy and Hematopoietic Stem Cell Transplant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE16Z17
Record Dates: First submitted 2017-12-15; First posted 2017-12-19 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Hematopoietic Stem Cell Transplant
Keywords: Music Therapy
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Therapy (Experimental): Participants in the experimental group will be given choices about how to proceed with the session: active or passive, improvisation, re-creative or receptive songs, or receptive (relaxation). Three music therapy sessions will be completed, the first within 24 hours of admission, the second 24-96 hours of session 1, and the final session the day before stem cell infusion.
  Interventions: Behavioral: Music Therapy
- No Music Therapy (Active Comparator): Participants randomized to the standard care group will be asked to rate the same symptoms as those in the experimental group. This will mark the beginning of a 45-minute control condition period during which the participants may fill the 45-minute time-period in whatever ways they choose.
  Interventions: Behavioral: No Music Therapy

INTERVENTIONS:
Behavioral: Music Therapy — No narcotic or anti-emetic therapy will be administered for at least 2 hours prior to music therapy session. Music therapy sessions will be administered by a board certified music therapist (MT-BC) and last approximately 45 minutes. Involvement in sessions will be based on therapist and patient availability.
  Arms: Music Therapy
Behavioral: No Music Therapy — Participants will fill the same 45 minute period in any way they choose; however, they will be asked to refrain from listening to recorded music during this time.
  Arms: No Music Therapy

SUMMARY:
The purpose of this randomized, controlled study is to determine the effects of pre-transplant music therapy on mood, distress, and physical functioning variables in patients undergoing Hematopoietic Stem Cell Transplant (HSCT).

DETAILED DESCRIPTION:
Primary Endpoint:

Compare the difference in distress via Distress Thermometer for patients who receive music therapy and those who do not.

Secondary Endpoints:

Compare the difference in patient perception of pain, anxiety, and mood via Numeric Rating Scale for patients who receive music therapy and those who do not.

Compare the difference in quality of life via Functional Assessment of Cancer Therapy-General (FACT-G7) for patients who receive music therapy and those who do not.

Compare the difference in the use of total narcotic medications in those who receive music therapy and those who do not (using morphine equivalent doses).

Study Design:

Participants randomized in the experimental group will receive a total of three sessions prior to stem cell infusion day. The first session will occur within 24 hours of admission to the bone marrow transplant (BMT) unit. The second session will occur between 24 - 96 hours after the first session, depending on transplant preparation regimen. The third session will occur on Day -1. For participants in the control group, assessments will be timed to emulate those in the experimental arm.

A decision tree for music therapy interventions will be employed in this study. Participants in the experimental group will be given choices about how to proceed with the session: active or passive, improvisation, re-creative or receptive songs, or receptive (relaxation).

Participants randomized to the standard care group will be asked to rate the same symptoms as those in the experimental group. This will mark the beginning of a 45-minute control condition period during which the participants may fill the 45-minute time-period in whatever ways they choose, however, they will be asked to refrain from listening to recorded music during this time. At the conclusion of 45-minutes, post-condition data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing inpatient allogeneic stem cell transplant
* Must be fluent in English
* Must be able to communicate verbally and have no significant hearing impairment
* Have capacity to provide consent
* All diagnosis, graft source, donor sources will be included.

Exclusion Criteria:

* Patients not meeting the above inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2019-06-21 (Actual)

PRIMARY OUTCOMES:
Change in Distress Score | From admission to day -1 (up to 9 days)
  Distress Thermometer assessments for both the experimental and standard care group will be given in the mid-late afternoon. This is an analog scale from 0-10 where 0 indicates no distress and 10 indicates extreme distress.

SECONDARY OUTCOMES:
Change in Pain Score | Within 24 hours of admission
  Before and after each music therapy session or control condition, participants will provide self-reported numeric ratings of pain/anxiety. The Numeric Rating Scale will be from 0-10, where 10 is the most pain/anxiety possible.
Change in Pain Score | Up to 96 hours after session 1 (120 hours from admission)
  Before and after each music therapy session or control condition, participants will provide self-reported numeric ratings of pain/anxiety. The Numeric Rating Scale will be from 0-10, where 10 is the most pain/anxiety possible.
Change in Pain Score | Up to 24 hours before procedure
  Before and after each music therapy session or control condition, participants will provide self-reported numeric ratings of pain/anxiety. The Numeric Rating Scale will be from 0-10, where 10 is the most pain/anxiety possible.
Change in Mood Score | Within 24 hours of admission
  Before and after each music therapy session or control condition, participants will report mood using the Rogers Happy/Sad Faces Scale, a five point visual analog scale.
Change in Mood Score | Up to 96 hours after session 1 (120 hours from admission)
  Before and after each music therapy session or control condition, participants will report mood using the Rogers Happy/Sad Faces Scale, a five point visual analog scale.
Change in Mood Score | Up to 24 hours before procedure
  Before and after each music therapy session or control condition, participants will report mood using the Rogers Happy/Sad Faces Scale, a five point visual analog scale.
Change in Quality of Life Score | From admission to day -1 (up to 9 days)
  The FACT-G7 is a seven-item assessment measuring cancer-specific quality of life. Seven items are scored on a 5-point scale (0-4), and patients are asked to indicate responses based on their experiences in the previous 7 days.
Total Narcotic Medication Use | From admission to day -1 (up to 9 days)
  Medication will be extracted from the electronic medical record and converted to morphine equivalent doses.

CONTACTS AND LOCATIONS:
Overall Officials: Navneet Majhail, MD, Principal Investigator — Cleveland Clinic, Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic, Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States